CLINICAL TRIAL: NCT03325569
Title: Reduced GLP-1 Response is Associated With Prediabetes in Women With Adverse Metabolic Phenotype of PCOS Independently of BMI
Brief Title: GLP-1 Response in Women With PCOS and Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, MD PhD, University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IGH PCOS and inkretins
Record Dates: First submitted 2017-10-24; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-06

CONDITIONS: Incretin Hormones in PCOS With Prediabetes
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NGT (Active Comparator): NGT - normal glucose tolerance. Women with PCOS and normal glucose tolerance
  Interventions: Diagnostic Test: oral glucose tolerance test
- IGH (Active Comparator): IGH - impaired glucose homeostasis Women with PCOS and impaired glucose homeostasis - that means impaired fasting glucose or impaired glucose tolerance.
  Interventions: Diagnostic Test: oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test — GLP1 response to oral glucose load during oral glucose tolerance test was assessed.

SUMMARY:
Women with PCOS are more prone to obesity which exacerbates insulin resistance, the abdominal fat disposition and metabolic risk of these patients. With development of obesity these women have high conversion rate from normal glucose tolerance to impaired glucose tolerance and in turn to type 2 diabetes.

Glucagon-like peptide 1 (GLP-1) is involved in body weight maintenance. Beside energy balance it is also involved in glucose homeostasis. Functional deficit in GLP-1 facilitates obesity. We investigated the link between the concentration of incretin hormones and glucose homeostasis, metabolic complications and the distribution of body composition in obese women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to menopause
* polycystic ovary sindrome (NICHD criteria)
* BMI of 30 kg/m2 or higher

Exclusion Criteria:

* type 1 or type 2 diabetes mellitus
* Cushing's syndrome or congenital (non-classic) adrenal hyperplasia
* personal or family history of MEN 2
* the use of medications known or suspected to affect reproductive or metabolic functions
* the use of statins within 90 days prior to study entery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
The main outcome was difference in fasting and after load GLP1 levels between two groups | 3h
  Patient GLP1 levels were measured at base point and in 120 min of 75-g OGTT. GLP1 levels were compared between groups

SECONDARY OUTCOMES:
The secondary outcome was to evaluate the between group difference in beta cell function, and visceral adipose tissue. | 3h
  At base point visceral adipose tissue (VAT) mass, volume and area were measured with DXA. To assess beta cell function static and dynamic parameters of beta cell function were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janez, MD PhD, Study Chair — University Medical Centre Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No